CLINICAL TRIAL: NCT03157258
Title: Social Network Intervention to Engage Community PLH to Engage in HIV Medical Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Yuri A. Amirkhanian, PhD, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO28750
Record Dates: First submitted 2017-05-09; First posted 2017-05-17 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2023-02

CONDITIONS: Human Immunodeficiency Virus; HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Network Endorsement (Experimental): All participants in this arm will receive two intervention elements: (1) they will receive a brief single care-related counseling session and referral to HIV medical care upon enrollment; and (2) all members of the HIV+ social networks will attend a multi-session group intervention during which they will be trained to deliver messages endorsing compliance with medical guidelines and adherence to medical treatment regimens to friends. Additionally, these leaders will be trained how to deliver effective messages.
  Interventions: Behavioral: Social Network Training
- HIV Counseling and Referral to Care (Active Comparator): All study participants will receive a brief single care-related counseling session and referral to HIV medical care at baseline.
  Interventions: Behavioral: Single Care-Related Counseling Session and Referral to Care

INTERVENTIONS:
Behavioral: Social Network Training — Members of HIV+ social networks randomized to this arm will be trained to endorse compliance with medical guidelines and adherence to medical treatment regimens to their friends.
  Arms: Social Network Endorsement
Behavioral: Single Care-Related Counseling Session and Referral to Care — Members of HIV+ social networks randomized to this arm will attend a single, brief care-related counseling session and referral to care at baseline.
  Arms: HIV Counseling and Referral to Care

SUMMARY:
People living with HIV infection (PLH) are clustered in friendship groups with other HIV+ persons, and an intervention delivered to all members of PLH social networks allows HIV+ people who are friends in day-to-day life to provide one another with support for entering, remaining, and adhering to HIV medical care. Moreover, an intervention delivered to groups attended by HIV+ persons who are friends increases HIV medical care engagement and decreases problem drinking more than individual counseling, probably because the network intervention harnessed mutual peer social support among friends who share the same HIV status, face similar coping issues, and interact together in day-to-day life. The planned research will be conducted in two phases in St. Petersburg, Russia.

DETAILED DESCRIPTION:
Phase I of the planned research will be the conduct of in-depth interviews with 30 HIV+ persons not in medical care or not adherent to anti-retroviral therapy (ART) regimens, including men and women representing diverse exposure risks (drug use, men who have sex with men, and heterosexual transmission). Interviews will elicit information on ways in which HIV-positive friends can support one another in HIV care entry, retention, and adherence; types of support from PLH friends that would best support treatment engagement; and how peer supports can lessen the negative effects of substance use on care engagement.

Phase 2 will recruit 48 out-of-care or ART nonadherent HIV+ individuals from community settings in St. Petersburg, Russia. These individuals, who are referred to as "network seeds," will invite their HIV+ friends, who will in turn invite their own HIV+ friends into the study, creating a sample of 48 networks (expected n=288, 6 members/network x 48 networks). Following baseline assessment of care engagement, ART adherence, treatment attitudes, psychosocial distress, substance use, and CD4+ and viral load, 24 networks (n=144 participants) will be randomized to an intervention condition and 24 networks (n=144) to the comparison condition. All members of each intervention condition network will together attend a 4-session intervention to strengthen attitudes, intentions, and skills for entering, remaining, and adhering to HIV medical care. Because participants will attend sessions with other individuals who are their own friends in day-to-day life, the intervention will build and increase mutual social support within each network for HIV care and adherence. Peer champions identified in each intervention network will attend 3 additional sessions in which they are guided to reinforce and help to sustain friends' medical care engagement. Intervention outcomes will be determined by baseline to 6- and 12-month followup change on primary measures of participant attendance at HIV medical care visits, adherence to ART regimens, and viral load as well as secondary measures of alcohol use, drug use, sexual risk behavior, treatment attitudes, and psychosocial distress.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older;
* Self-report as being HIV-positive, with positive HIV status confirmed in study-provided testing;
* Except for initial seeds, must be named by an already-enrolled participant as a PLH friend; and
* Do not plan to move from the St. Petersburg, Russia, area for the next 18 months.

Exclusion Criteria:

* Age 17 or younger;
* Self-report as HIV-negative or HIV-positive serostatus is not confirmed by testing;
* Not be named as a PLH friend by an already-enrolled participant; and
* Intend to move from the St. Petersburg, Russia, area during the next 18 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
HIV viral load values | 0 months; 6 months; 12 months
  Change in HIV viral load values at baseline will be compared with HIV viral load values determined at 6 months post-intervention and 12 months post-intervention.
HIV medical care visits | 0 months; 6 months; 12 months
  Change in the number of self-reported HIV medical care visits during the prior six months, comparing the number of visits reported at baseline to the number reported at six and twelve months at post-intervention followup assessments.
Antiretroviral medication adherence | 0 months; 6 months; 12 months
  Change in medication adherence during the past 30 days (as measured by the visual analogue scale; J.C. Walsh, et al, 2002), comparing the adherence percentage reported at baseline to the adherence percentage reported at the six and twelve month postintervention followup assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Yuri A. Amirkhanian, PhD, Principal Investigator — Medical College of Wisconsin; Jeffrey A. Kelly, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No